CLINICAL TRIAL: NCT06005779
Title: An Ambispective Cohort Study on the Prognosis and Its Influencing Factors of Borderline Personality Disorder
Brief Title: A Study on the Outcome and Its Influencing Factors in Patients With Borderline Personality Disorder
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Wuhan Mental Health Centre (Other)
Responsible Party: Sponsor
Other Study IDs: KY2018.77
Record Dates: First submitted 2023-08-15; First posted 2023-08-22 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Borderline Personality Disorder
MeSH Terms: conditions — Borderline Personality Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Borderline personality disorder (BPD) is a difficult chronic mental illness. This diagnosis is common in Western countries. Our researchers want to study the outcome and its influencing factors of BPD for the first time in China. Patients with BPD who had been hospitalized in Wuhan Mental Health Center were selected as the subjects. The researchers retrospectively collected the most recent hospitalization data of these patients, and then prospectively follow up them for 2 years to see how their condition will change. By analyzing all data, researchers hope to know deeply about the development law of this illness, and to provide evidence for releasing these patients' suffering.

DETAILED DESCRIPTION:
This study is an ambispective cohort study. The information collected in the retrospective part mainly included demographic data, comorbid psychiatric diagnosis, psychotherapeutive and pharmacotherapeutive data, times of hospitalization and patients' contact information. The above data were derived from electronic medical records. After informed consent, prospective follow-up was initiated primarily by telephone interviews and web-based questionnaires, or by in-person assessments at hospital return visits. Enrolled patients will be followed up at 6-month intervals after the first follow-up to assess psychiatric diagnosis, social function, and quality of life. The researchers are senior psychiatrists, all of whom received training on the use of questionnaires and inter-investigator consistency before the follow-up.

Cox Proportional Hazard Model is used to analyze the influencing factors of remission of BPD, and Generalized Estimating Equation Model is used to analyze the influencing factors of the patients' social function and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of BPD based on ICD-10 (F60.3)

Exclusion Criteria:

* Comorbidity with severe physical disease
* Comorbidity with neurological diseases such as epilepsy
* Comorbidity with mental retardation

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Inpatients at the Wuhan Mental Health Center
Sampling Method: Non-Probability Sample
Enrollment: 270 (Estimated)
Dates: Start 2021-10-22 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
remission rate | After the first follow-up, patients will be followed up every 6 months, and the total follow-up time was 2 years.
  The remission rate is calculated as the number of patients who no longer met the diagnostic criteria for BPD for at least 6 months divided by the total number of enrolled patients. The diagnostic tool is ICD-10 (F60.3).

SECONDARY OUTCOMES:
social disability | After the first follow-up, patients will be followed up every 6 months, and the total follow-up time was 2 years.
  Social disability refers to the patient's occupation, family, social life, personal life and other aspects of functional deficits, using Social Disability Screening Schedule (SDSS) to assess.
quality of life | After the first follow-up, patients will be followed up every 6 months, and the total follow-up time was 2 years.
  Someone's quality of life is the extent to which their life is comfortable or satisfying. The study used WHOQOL-BREF to assess patients' quality of life in the physical, psychological, social relationship, and environmental domains.

CONTACTS AND LOCATIONS:
Overall Officials: Fan Yang, Master, Study Director — Wuhan Mental Health Centre
Locations (1):
- Wuhan Mental Health Centre, Wuhan, Hubei, China